CLINICAL TRIAL: NCT03974698
Title: Uncemented Hemiarthroplasty, Radiological Features Comparing Lateral Versus Anterolateral Approach: A Follow-up of a Randomized Controlled Trial.
Brief Title: Uncemented Hemiarthroplasty, Radiological Features Comparing Lateral Versus Anterolateral Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Raymond Tellefsen
Record Dates: First submitted 2019-05-27; First posted 2019-06-05 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2019-05

CONDITIONS: Femoral Neck Fractures; Hemiarthroplasty; Heterotopic Ossification
Keywords: femoral offset; leg length discrepancy; valgus/varus position; Lateral approach; Anterolateral approach
MeSH Terms: conditions — Femoral Neck Fractures; Ossification, Heterotopic; Leg Length Inequality; Genu Valgum | interventions — Hemiarthroplasty

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants attempted masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterolateral approach (Active Comparator): Standard x-ray on all operated patients was taken pre- and postoperative and at 3 and 12 moths. Including an AP pelvis and lateral view of the hip.
  Interventions: Procedure: Hemiarthroplasty
- Lateral approach (Active Comparator): Standard x-ray on all operated patients was taken pre- and postoperative and at 3 and 12 moths. Including an AP pelvis and lateral view of the hip.
  Interventions: Procedure: Hemiarthroplasty

INTERVENTIONS:
Procedure: Hemiarthroplasty — Radiological features comparing the femoral stem position is measured on the postoperative x-ray. Presence of heterotopic ossification is assessed on the 12 months follow up.

SUMMARY:
Uncemented Hemiarthroplasty, Radiological Features Comparing Lateral Versus Anterolateral Approach. Comparing leg length discrepancy, femoral offset, valgus/varus position of the stem. Also is there a difference in heterotopic ossification at 12 months.

DETAILED DESCRIPTION:
Between January 2014 and July 2017 a RCT was conducted at Sorlandet Hospital Kristiansand, Norway. The trial was approved by the regional ethics committee (2013/1853/REK) and registered at ClinicalTrials.gov (ClinicalTrials.gov Identifier NCT02028468). This study is a follow-up on the same study population.

150 patients (70 to 90 years) with a displaced femoral neck fracture was randomized to be operated With either anterolateral og Direct lateral surgical approach. Investigators want to compare the radiological features of the femoral stem between the two Groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 70 and 90 years of age with displaced femoral neck fractures
* Intact cognitive function
* Ability to walk with or without a walking aid prior to falling.

Exclusion Criteria:

* Dementia
* Fractures in pathologic bone
* Patients not belonging to the hospital community
* Patients with sepsis or local infection
* Fracture not eligible to be treated with a hemiarthroplasty

Ages: 70 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Leg length | Immediately after surgery
  The perpendicular distance between a horizontal line passing through the lower edge of the teardrop to the ipsilateral center of the femoral head

SECONDARY OUTCOMES:
Femoral offset | Immediately after surgery
  The distance between the longitudinal axis of the femur to the centre of the femoral head and the distance from the centre of the femoral head to a perpendicular line passing through the medial edge of the teardrop
Valgus/varus stem position | Immediately after surgery
  Stem position in relation to the femoral axis
Heterotopic ossification | 1 year
  Classified as type 1-4 according to Brooker classification
Canal fill ratio | Immediately after surgery
  Was evaluated at the following points; 2 cm above the lower trochanter, at the tip of the lower trochanter, 2 cm and 7 cm below the tip of lesser trochanter

OTHER OUTCOMES:
Canal Flare index | Immediately after surgery
  the ratio of the intracortical width of the femur at 20 mm proximal to the tip of lesser trochanter and isthmus at 10 cm distally
Dorr classification | Immediately after surgery
  Morphology of the proximal femur
Cortical Thickness Index | Immediately after surgery
  the ratio of cortical width minus endosteal width, to cortical width at 10 cm below the tip of lesser trochanter

CONTACTS AND LOCATIONS:
Overall Officials: Lars Nordsletten, Prof, Principal Investigator — Oslo University Hospital
Locations (1):
- Sorlandet Hospital, Kristiansand, Norway

REFERENCES:
- [Background] Ugland TO, Haugeberg G, Svenningsen S, Ugland SH, Berg OH, Hugo Pripp A, Nordsletten L. Less periprosthetic bone loss following the anterolateral approach to the hip compared with the direct lateral approach. Acta Orthop. 2018 Feb;89(1):23-28. doi: 10.1080/17453674.2017.1387730. Epub 2017 Oct 17. PMID 29037093
- [Background] Ugland TO, Haugeberg G, Svenningsen S, Ugland SH, Berg OH, Pripp AH, Nordsletten L. Biomarkers of muscle damage increased in anterolateral compared to direct lateral approach to the hip in hemiarthroplasty: no correlation with clinical outcome : Short-term analysis of secondary outcomes from a randomized clinical trial in patients with a displaced femoral neck fracture. Osteoporos Int. 2018 Aug;29(8):1853-1860. doi: 10.1007/s00198-018-4557-y. Epub 2018 May 22. PMID 29789919
- [Derived] Tellefsen RA, Ugland T, Bjorndal MM, Ugland S, Pripp AH, Nordsletten L. Increased risk of high-grade heterotopic ossification using direct lateral approach versus a muscle-sparing anterolateral approach to the hip: radiological results from a randomised trial in patients with a femoral neck fracture treated with hemiarthroplasty. Hip Int. 2023 Jul;33(4):789-796. doi: 10.1177/11207000221097639. Epub 2022 May 18. PMID 35585787

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/98/NCT03974698/Prot_SAP_000.pdf